CLINICAL TRIAL: NCT03025373
Title: Virtual Reality Stimulation to Enhance Cognitive Function of Intensive Care Unit Patients
Status: Completed | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: University of Bern (Other)
Responsible Party: Sponsor
Other Study IDs: 2016-01652
Record Dates: First submitted 2017-01-16; First posted 2017-01-19 (Estimated); Last update posted 2019-05-03 (Actual); Status verified 2019-05

CONDITIONS: Cognitive Impairment, Mild; Quality of Life
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients - prolonged ICU stay (> 5 days): Controlled visual and acoustic stimulation in a virtual reality setting
  Interventions: Other: Visuo-acoustic stimulation
- Heart surgery patients (< 5 days): Controlled visual and acoustic stimulation in a virtual reality setting
  Interventions: Other: Visuo-acoustic stimulation

INTERVENTIONS:
Other: Visuo-acoustic stimulation — Controlled visual and acoustic stimulation in a virtual reality setting

SUMMARY:
An observational study will be conducted in the ICU (Intensive care unit) including patients with heart surgery (< 5 days) and prolonged ICU stay (> 5 days). Patients will receive 5 min Virtual reality stimulation per day. A modified version of the Oculus Rift VR glasses (Facebook inc., USA) with stereoscopic vision and stereo sound will be used to present the virtual world to patients. An integrated eye tracker will measure oculomotor responses that will be synchronized with the physiological data recording. All participants will undergo neuropsychological testing after ICU stay, and after a three-months follow-up. Quality of life prior to the ICU stay will be enquired from relatives. Main outcome variable is the explorative behaviour (attention). Secondary outcomes are the quality of life and cognitive functioning.

ELIGIBILITY:
Inclusion Criteria:

* Age > =18
* Speak German or French
* Are able to participate the follow up measurements
* Written informed consent

Exclusion Criteria:

* Visual impairments
* Cognitive impairments
* Cognitive impairments
* Craniocerebral injury before admitting the ICU
* Already admitted the intensive care unit (last year) or at reentry
* Psychotic disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population consist of adults on the intensive care unit
Sampling Method: Non-Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2019-04-01 (Actual)

PRIMARY OUTCOMES:
Attention measurement in patients in the intensive care unit | Changes from baseline in attention measurement during and after admission (3 Month) to the ICU
  The attention is measured via explorative behaviour of the subject. This means an eye tracker is used to measure eye movements, fixation duration and number of fixations, which can be used to calculate the explorative behaviour.

SECONDARY OUTCOMES:
Quality of Life | After 3 months after admission to the ICU
  The quality of life are examined via EuroQol (EQ-5D-5L) questionnaire
Cognitive functioning | Changes from baseline in cognitive functioning measurement after admission (3 Month) to the ICU
  The cognitive abilities are examined via CERAD test battery (Consortium to Establish a Registry for Alzheimer's Disease) this includes word fluidity, Boston Naming Test (BNT), mini-mental state examination (MMSE), word list memory, constructive practice, word list retrieve, word list recognition, constructive practice (retrieve)

CONTACTS AND LOCATIONS:
Overall Officials: Marie- Madlen Jeitziner, Dr., Study Chair — University hospital of Bern
Locations (1):
- Universitätsklinik für Intensivmedizin, Inselspital, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brummel NE, Jackson JC, Girard TD, Pandharipande PP, Schiro E, Work B, Pun BT, Boehm L, Gill TM, Ely EW. A combined early cognitive and physical rehabilitation program for people who are critically ill: the activity and cognitive therapy in the intensive care unit (ACT-ICU) trial. Phys Ther. 2012 Dec;92(12):1580-92. doi: 10.2522/ptj.20110414. Epub 2012 May 10. PMID 22577067
- [Background] Brummel NE, Girard TD, Ely EW, Pandharipande PP, Morandi A, Hughes CG, Graves AJ, Shintani A, Murphy E, Work B, Pun BT, Boehm L, Gill TM, Dittus RS, Jackson JC. Feasibility and safety of early combined cognitive and physical therapy for critically ill medical and surgical patients: the Activity and Cognitive Therapy in ICU (ACT-ICU) trial. Intensive Care Med. 2014 Mar;40(3):370-9. doi: 10.1007/s00134-013-3136-0. Epub 2013 Nov 21. PMID 24257969
- [Background] Cutler LR, Hayter M, Ryan T. A critical review and synthesis of qualitative research on patient experiences of critical illness. Intensive Crit Care Nurs. 2013 Jun;29(3):147-57. doi: 10.1016/j.iccn.2012.12.001. Epub 2013 Jan 9. PMID 23312486
- [Background] Jackson JC, Ely EW. Cognitive impairment after critical illness: etiologies, risk factors, and future directions. Semin Respir Crit Care Med. 2013 Apr;34(2):216-22. doi: 10.1055/s-0033-1342984. Epub 2013 May 28. PMID 23716312
- [Background] Luke SG, Henderson JM. The Influence of Content Meaningfulness on Eye Movements across Tasks: Evidence from Scene Viewing and Reading. Front Psychol. 2016 Mar 1;7:257. doi: 10.3389/fpsyg.2016.00257. eCollection 2016. PMID 26973561
- [Background] Needham DM, Dinglas VD, Bienvenu OJ, Colantuoni E, Wozniak AW, Rice TW, Hopkins RO; NIH NHLBI ARDS Network. One year outcomes in patients with acute lung injury randomised to initial trophic or full enteral feeding: prospective follow-up of EDEN randomised trial. BMJ. 2013 Mar 19;346:f1532. doi: 10.1136/bmj.f1532. PMID 23512759
- [Background] Pandharipande PP, Girard TD, Jackson JC, Morandi A, Thompson JL, Pun BT, Brummel NE, Hughes CG, Vasilevskis EE, Shintani AK, Moons KG, Geevarghese SK, Canonico A, Hopkins RO, Bernard GR, Dittus RS, Ely EW; BRAIN-ICU Study Investigators. Long-term cognitive impairment after critical illness. N Engl J Med. 2013 Oct 3;369(14):1306-16. doi: 10.1056/NEJMoa1301372. PMID 24088092
- [Background] Wolters AE, Slooter AJ, van der Kooi AW, van Dijk D. Cognitive impairment after intensive care unit admission: a systematic review. Intensive Care Med. 2013 Mar;39(3):376-86. doi: 10.1007/s00134-012-2784-9. Epub 2013 Jan 18. PMID 23328935